CLINICAL TRIAL: NCT02019862
Title: TRJ PMCF Köln: 2-years Results
Brief Title: TRJ Post Market Clinical Follow Up
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1314
Record Dates: First submitted 2013-12-04; First posted 2013-12-24 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Total Hip Arthroplasty
Keywords: Total hip arthroplasty; TRJ; PMCF; Hip stem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TRJ®
  Interventions: Device: TRJ® Total Hip Arthroplasty

INTERVENTIONS:
Device: TRJ® Total Hip Arthroplasty

SUMMARY:
Clinical and radiological 2 years results of TRJ® Hip Stem.

ELIGIBILITY:
Inclusion:

* TRJ® implantation performed
* patient consent available for participation in the study

Exclusion:

* permanent cortisone therapy
* alcohol or drug abuse

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: specialist clinical centre
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Implant Survival | 24 months

SECONDARY OUTCOMES:
Clinical Outcome | 24 months
  Harris Hip Score
Osteolysis | 24 months
  Radiological Outcome
Ossification | 24 months
  Radiological Outcome
Migration | 24 months
  Radiological Outcome
TRJ® Implant Position | 24 months
  Radiological Outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Dreifaltigkeitskrankenhaus Köln, Cologne, Germany